CLINICAL TRIAL: NCT04778995
Title: The Scientific and Technological Research Council of Turkey
Brief Title: Online Training Program Model for Effective Management of Nursing Services in Times of Crisis Such as Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Handan Alan, Assistant Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-90
Record Dates: First submitted 2021-01-20; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Pandemics; Crisis State; Nursing; Education
Keywords: Online Training Program; Nursing Management; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manager nurses (Experimental group) (Experimental): Manager nurses who participated in the structured training program based on qualitative data. Web based training program was the intervention for this group.
  Interventions: Other: Structured online training program for effective management of nursing services
- Manager nurses (Control group) (No Intervention): Manager nurses who were not included to the structured training program based on qualitative data. No intervention was performed for this group.

INTERVENTIONS:
Other: Structured online training program for effective management of nursing services — An online structured training program was prepared to reach out to manager nurses for increasing their knowledge regarding the effective management of nursing services in crisis periods. A web page was structured with the support of a professional computer engineer.
  Participant manager nurses could log into the system via a personal username and password on the main login screen of the site. In this page, there is an "Informed Consent Form".
  In the "Download Training Documents" link; the educational content prepared in sections was presented. Educational content consisted of the issues such as: Management of Crises and Emergency Situations, Leadership in Crisis, Planning and Managing Nurse Human Power in Crisis, Supervision and Management of Patient Care, Logistics and Support Services, Communication in Extraordinary Situations, Motivation Tools Used in Extraordinary Situations, Stress Management During Crisis and Employee Adaptation and Training in Crisis.
  Arms: Manager nurses (Experimental group)

SUMMARY:
This project is designed to determine the experiences of nurses working in healthcare organizations in the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic and their approaches to problems experienced in qualitative design and from these results, a web-based education model is prepared for the effective management of nursing services, to increase the knowledge and skills of manager nurses. It was carried out in a quasi-experimental design.

In the qualitative phase of the study, 28 people nurses were included (14 manager nurses and 14 nurses), and 61 nurse managers, including 30 intervention and 31 control group, participated in the randomized controlled quasi-experimental quantitative phase. Qualitative data were analyzed using the "Interview Form" through an in-depth interview method; Experimental data were collected via a pre- and post-questionnaire from nine web-based training videos. Qualitative data were analyzed in the MAXQDA 2020 program, and experimental data were analyzed in the Statistical Package for the Social Sciences (SPSS) 21.0 package program.

Findings obtained from the qualitative stage; The problems regarding the institution's general management, the problems and approaches experienced by the nurses, and the problems and approaches experienced by the manager nurses were evaluated under three main themes. A pre-test / post-test questionnaire was applied to the intervention and control groups created due to the analysis of qualitative data.

DETAILED DESCRIPTION:
Purpose and Type of the Research This stage was conducted as a randomized controlled quasi-experimental study to evaluate web-based education's effect on the effective management of nursing services during the SARS-CoV-2 pandemic and similar crisis periods.

Place and Time of the Study The research was conducted with executive nurses working in public and private hospitals serving as the SARS-CoV-2 pandemic hospital in Istanbul between October 15 and November 30, 2020.

Study Population and Sample The study's universe was composed of the members of Association of Nurse Managers and those who returned after the announcement, working as a nurse manager in Istanbul. The sampling of the study included manager nurses who met the inclusion criteria with the purposeful sampling method.

Determination of Intervention and Control Groups: Randomization Association of Nurse Managers members were asked whether they would like to participate in the study by e-mail. An online introductory information form link was sent to the members who stated they would like to participate. A number was given to the members according to the order they filled out this form, and randomization was carried out after this process.

It is the determination of the randomization intervention group in which the group at the beginning of the study will be examined completely randomly. Randomization was performed to provide an equal number of samples in the intervention and control groups and ensure that both groups were similar in terms of all factors except the website, whose effectiveness will be examined. "Simple randomization method" was chosen as the randomization method to provide an equal number of samples in two groups. Randomization was performed using the website https://www.randomizer.org/ in a computer environment. Participants were divided into intervention or control groups according to randomization results. An application flow chart was prepared using the CONSORT chart.

Data Collection Tools The data were collected by participant information form, pre-test, and post-test.

Participant information form: The form prepared by the researcher's questions the participants' personal and professional characteristics. In the personal characteristics section of the form, there are seven questions, namely name-surname, e-mail address, gender, age, marital status, educational status, the field of graduate education; In the occupational characteristics section, there are five questions, namely, the status of the institution and institution being a fully pandemic hospital, position, professional experience, and management experience.

Pre-test / Post-test: Before preparing web-based training videos, 2 questions were asked by our expert trainers who came to the training about the subjects they will tell. These multiple-choice questions have five options, and the participants try to find the correct answer.

Preparation of the Website Preparation of Website Content Website; It was prepared to increase manager nurses' knowledge needs regarding the effective management of nursing services in crisis periods. A web page named "Executive Nurse Training Program" was created with the support of a computer engineer for the website's design.

On the main login screen of the site page created, an area has been created where they can log into the system by using a personal user name and password. In this area, under the "I accept the Terms and Conditions" tab, there is an "Informed Consent Form". It is not possible to register to the system before this section is approved. It is necessary to use the username and password for every new login to the system. On the main page; Along with the expression welcome to the training program, short information and video explaining the purpose of the program are available. Towards the bottom of the page; There are explanations about the process in which The Scientific and Technological Research Council of Turkey supports the project. At the bottom of the page, there is the section where the names and surnames of the project team and the institution they work for and the project e-mail address for communication. In the "Educators" button, the expert educators' resumes who support our project can be accessed in the training videos. In the "Download Training Documents" link; The educational content prepared in sections was presented. Educational content; "Management of Crises and Emergency Situations," "Leadership in Crisis," "Planning and Managing Nurse Human Power in Crisis," "Supervision and Management of Patient Care," "Logistics and Support Services," "Communication in Extraordinary Situations," "Motivation Tools Used in Extraordinary Situations," "Stress Management During Crisis "and" Employee Adaptation and Training in Crisis. " Preparation of Training Videos In line with the data obtained from the interviews at the first stage of the study, the training titles were determined following the literature. To make presentations in the determined educational titles, the researchers determined experts in their fields with a common opinion. The people determined for the training were contacted. The researchers were given appointments at the appropriate day and time. The video footage was made by researchers and scholarship students in the classroom allocated by the Dean's Office of Florence Nightingale Nursing Faculty. Video shootings were made by paying attention to social distance rules. After the shooting, the trainers watched videos, and their approval was obtained. In some of the training videos, the videos were retaken because they frequently paused and used the expressions "like" frequently. After the filming was completed, the videos were edited by the research director and scholarship students. The training videos were shared with all researchers before they were uploaded to the web page, and a final check was made.

Collection of Data The application of the research was carried out in two steps. Web-based training was given to the manager nurses, who accepted to participate in the study and incidentally joined the intervention group between 15 October and 30 November 2020. Manager nurses have accessed the site's home page and training content with their unique username and password via the designated website. Manager nurses were able to access the training content from their mobile phones, tablets, or computers using any internet connection, in any place and the time frame they wanted. To open the educational content prepared in the form of a video, they had to solve the "pre-test." The manager nurses were informed that they can access the training content in any time period they want between October 15 and November 30, 2020 but will not access the program when the specified time is over. Therefore, reminder messages were sent via e-mail to those who did not watch training videos for a long time. Manager nurses completed the training content according to their own programs. When they felt sufficient about the training content and wanted to terminate the training, they were made to complete the training by solving the "final test." After the training was completed, a "Participation Certificate" was sent to the manager nurses via e-mail.

Manager nurses completed the training content according to their own programs. When they felt sufficient about the training content and wanted to terminate the training, they were made to complete the training by solving the "final test." After the training was completed, a "Participation Certificate" was sent to the manager nurses via e-mail.

The manager nurses who accepted to participate in the study were asked to complete the online pre-test sent on the link by explaining that no intervention was applied to the control group. They were included in the control group via e-mail between 15-25 October 2020. Participants who took the pre-test were sent a post-test link via e-mail between 1-10 December. In the follow-up of the application made to the intervention group, while the intervention group participants answered the final test, the manager nurses in the control group were also provided with the final test. Then, the web address was made available so that the control group participants could access the training contents. The control group participants were created a new password and username, and the necessary explanations were sent by e-mail to enable them to participate in the training, and a "Participation Certificate" was sent to the participants who finished.

Ethical Aspect of the Research Ethics committee approval was obtained from Istanbul University-Cerrahpasa Social and Human Sciences Research Ethics Committee for the research. Written permission was obtained from Association of Nurse Managers board members. Verbal and written information about the study was given to the individuals who met the inclusion criteria in the study and written informed consent of the patients who accepted it was obtained. It was stated that the information obtained at the end of the research would not be used anywhere other than the research report and scientific publications to be produced from the project and that individuals can leave the research at any time.

ELIGIBILITY:
Inclusion Criteria:

* Preferably being a member of Association of Nurse Managers,
* Being a manager nurse,
* To be a manager for at least two years,
* To be at least a bachelor's degree,
* Working,
* It is to volunteer to participate in the study.

Exclusion Criteria:

* Participating in the first stage of the research,
* Not being an executive nurse,
* Less than two years of management experience
* To be a high school or associate degree graduate,
* Not working actively,
* Not willing to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change after online training program on the management of nursing services in times of crisis | Two months
  While a statistically significant change is expected between the pre-test and post-test scores of the experimental group, no statistically significant change is expected between the pre-test and post-test scores of the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Veenema TG, Deruggiero K, Losinski S, Barnett D. Hospital Administration and Nursing Leadership in Disasters: An Exploratory Study Using Concept Mapping. Nurs Adm Q. 2017 Apr/Jun;41(2):151-163. doi: 10.1097/NAQ.0000000000000224. PMID 28263273
- [Result] Wang H, Feng J, Shao L, Wei J, Wang X, Xu X, Shao R, Zhang M, He J, Zhao X, Liang T. Contingency management strategies of the Nursing Department in centralized rescue of patients with coronavirus disease 2019. Int J Nurs Sci. 2020 Apr 4;7(2):139-142. doi: 10.1016/j.ijnss.2020.04.001. eCollection 2020 Apr 10. PMID 32292636
- [Result] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538